CLINICAL TRIAL: NCT03518047
Title: Risankizumab Versus Placebo in a Randomized, Double Blind, Parallel Group Trial in Moderate to Severe Plaque Psoriasis to Assess Safety and Efficacy After 16 Weeks of Treatment in the Russian Federation (IMMpress)
Brief Title: Risankizumab Therapy Versus Placebo for Subjects With Psoriasis in the Russian Federation
Acronym: IMMPRESS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M16-176
Record Dates: First submitted 2018-05-04; First posted 2018-05-08 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Psoriasis
Keywords: Plaque Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — risankizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo for risankizumab by subcutaneous (SC) injection.
  Interventions: Drug: placebo for rizankizumab
- Risankizumab (Experimental): Risankizumab by subcutaneous (SC) injection.
  Interventions: Drug: risankizumab

INTERVENTIONS:
Drug: risankizumab — rizankizumab subcutaneous (SC) infusion
  Other Names: ABBV-066; BI 655066
  Arms: Risankizumab
Drug: placebo for rizankizumab — placebo for rizankizumab subcutaneous (SC) infusion
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of risankizumab compared to placebo in subjects with moderate to severe chronic plaque psoriasis in the Russian Federation.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of chronic plaque psoriasis (with or without psoriatic arthritis) for at least 6 months before the first administration of study drug.
* Moderate to severe chronic plaque psoriasis at both Screening and Baseline (Randomization) Visits
* Candidates for systemic therapy or phototherapy for psoriasis treatment as assessed by the investigator

Exclusion Criteria:

* Prior therapy with an anti-interleukin (IL)-17 or anti-IL12/23p40 or anti-IL-23p19 inhibitor
* Concurrent therapy with a biologic and/or other systemic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2020-02-11 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with a 90% reduction from Baseline Psoriasis Area and Severity Index (PASI 90) at Week 16 | Week 16
  The PASI score is an established measure of clinical efficacy for psoriasis medications.

SECONDARY OUTCOMES:
Proportion of participants with Static Physician Global Assessment (sPGA) score of clear or almost clear (0, 1) at Week 16 | Week 16
  The sPGA is based on the physician's assessment of the average thickness, erythema, and scaling of all psoriatic lesions.
Proportion of participants with a 75% reduction from Baseline Psoriasis Area and Severity Index (PASI 75) at Week 16 | Week 16
  The PASI score is an established measure of clinical efficacy for psoriasis medications.
Proportion of participants with a 100% reduction from Baseline Psoriasis Area and Severity Index (PASI 100) at Week 16 | Week 16
  The PASI score is an established measure of clinical efficacy for psoriasis medications.
Proportion of Participants Achieving a Dermatology Life Quality Index (DLQI) Score of 0 or 1 at Week 16 | Week 16
  The DLQI is a self-administered, ten-question questionnaire used to assess the effect of different skin diseases on a subject's quality of life, overall health, and disability status. Scores range from 0 (not relevant/not at all) to 3 (very much).

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (6):
- Russia (6):
  - GBUZ Clinical Dermatovenerology Dispensary of MoH of Krasnodar region /ID# 201713, Krasnodar, Krasnodarskiy Kray
  - Family Outpatient clinic#4 LLC /ID# 207441, Korolev, Moscow
  - SBHI KVD # 10 Clinic of Dermatology and venerology /ID# 200615, Saint Petersburg, Sankt-Peterburg
  - LLC ArsVitae Severo-Zapad /ID# 200658, Saint Petersburg, Sankt-Peterburg
  - LLC Kurator /ID# 200616, Saint Petersburg, Sankt-Peterburg
  - Alliance Biomedical Ural Group /ID# 201681, Izhevsk, Udmurtiya Republic

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Odnopozova L, Edin A, Sukharev A, Wu T, Aydin K, Kelly M, Khotko A. Risankizumab for the Treatment of Moderate to Severe Plaque Psoriasis in the Russian Federation. Dermatol Ther (Heidelb). 2022 Sep;12(9):2063-2075. doi: 10.1007/s13555-022-00776-0. Epub 2022 Aug 2. PMID 35917057
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/clinical-trials/risankizumab_M16-176.pdf